CLINICAL TRIAL: NCT00398177
Title: Clinical and Pathologic Studies in Non-Hodgkin's Lymphoma and Hodgkin's Disease
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Biospect Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LYM0001; 76973 (Other: Stanford University Alternate IRB Approval Number); LYM0001 (Other: OnCore); IRB-13500 (Other: Stanford IRB)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin's Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tumor tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize the molecular and cell biology of the tumor cells in lymphoma.

DETAILED DESCRIPTION:
This research involves the study of lymphoma cells in order to better understand how the disease grows and spreads. This study may lead to the development of special materials that could be used, in the future, to treat lymphoma or to follow the response of lymphoma to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hodgkin's disease or non-Hodgkin's lymphoma, any cellular classification, any stage, any grade.
* Adult or pediatric patients receiving lymph node excision for purposes other than cancer therapy (i.e. tonsillectomy, sleep apnea).
* A routine procedure for tissue collection is planned.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients without NHL or Hodgkin's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any type of NHL or Hodgkin's disease.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 1999-01; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
Collection of tumor tissue to characterize the molecular and cell biology of tumor cells in lymphoma. | The study will continue indefinitely.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Roschewski M, Kurtz DM, Westin JR, Lynch RC, Gopal AK, Alig SK, Sworder BJ, Cherng HJ, Kuffer C, Blair D, Brown K, Goldstein JS, Schultz A, Close S, Chabon JJ, Diehn M, Wilson WH, Alizadeh AA. Remission Assessment by Circulating Tumor DNA in Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec;43(34):3652-3661. doi: 10.1200/JCO-25-01534. Epub 2025 Aug 13. PMID 40802906
- [Derived] Kurtz DM, Scherer F, Jin MC, Soo J, Craig AFM, Esfahani MS, Chabon JJ, Stehr H, Liu CL, Tibshirani R, Maeda LS, Gupta NK, Khodadoust MS, Advani RH, Levy R, Newman AM, Duhrsen U, Huttmann A, Meignan M, Casasnovas RO, Westin JR, Roschewski M, Wilson WH, Gaidano G, Rossi D, Diehn M, Alizadeh AA. Circulating Tumor DNA Measurements As Early Outcome Predictors in Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2018 Oct 1;36(28):2845-2853. doi: 10.1200/JCO.2018.78.5246. Epub 2018 Aug 20. PMID 30125215